CLINICAL TRIAL: NCT01357928
Title: Procedure for the Reference Range Study for Haemoscope Reagents
Brief Title: Thromboelastography (TEG) Reference Range Study
Status: Completed | Type: Observational
Sponsor: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CLN-100048C
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Coagulation
Keywords: TEG; Thromboelastography; Coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers

SUMMARY:
As part of a system wide reagent verification plan Haemoscope Corporation will be running a study to verify the reference intervals of many of the reagents. Reference intervals will be constructed following the guidelines set out in CLSI document C28-A3c. This guideline calls for a reference interval to be constructed from at least 120 donors. Some reagents currently have ranges in place based on fewer donors than that stated in the guideline. This procedure will provide additional testing results to meet the requirements outlined in the CLSI guideline. Reagents that currently have no reference intervals will be tested and will include a minimum of 146 donors.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over the age of 18 years.

Exclusion Criteria:

* Genetic bleeding disorders
* Currently Pregnant
* Oral Contraceptives
* On anti-coagulants or anti-platelet therapy
* Took ASA (Acetylsalicylic Acid)within 1 week prior
* Recent surgery (within 4 weeks)
* Recent injury leading to substantial bruising (within 2 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William A Heaton, M.D., Principal Investigator — NSLIJ Health System
Locations (1):
- North Shore-Long Island Jewish Health System, Manhasset, New York, United States